### INVESTIGATOR-INITIATED STUDY PROPOSAL

# A Prospective Evaluation of Tissue Sealant to Prevent Epithelial Ingrowth in Repeat LASIK Surgery

The following is an investigator initiated study proposal to evaluate the relative effectiveness of the ReSure® Sealant at preventing epithelial ingrowth after LASIK flap re-lift.

Principle Investigator: Edward E. Manche, MD

**Funding:** Ocular Therapeutix, Inc. – \$ gift. SPO pending.

#### Introduction

It is well-known that a small percentage of patients will have epithelial ingrowth after primary LASIK and that preoperative refractive error is a correlated factor. The effects of that ingrowth can be glare and halos; ingrowth is a significant cause of dissatisfaction after LASIK. The incidence of epithelial ingrowth is significantly higher after flap re-lift for treatment of residual refractive error. It has been hypothesized that cell migration into the flap/cornea interface postoperatively is a primary reason for such ingrowth. A sealed interface may therefore have some utility in preventing epithelial ingrowth after flap re-lift.

The following investigator-initiated study proposal is designed to determine if a lower-than-typical rate of epithelial ingrowth occurs when a LASIK flap re-lift is performed and the replaced flap is sealed with ReSure sealant.

**Study specific aims:** Tissue sealant has been effectively used to prevent recurrence of epithelial ingrowth under the LASIK flap. The aim of the study is to see if tissue sealant can be used to prevent epithelial ingrowth from occurring in the first place. This would allow for patients to undergo LASIK flap lift surgery with greater safety.

**Unpublished data:** There is no unpublished data on the prophylactic use of tissue sealant to prevent the occurrence of epithelial ingrowth under the flap. It has been used successfully to prevent recurrence of epithelial ingrowth under the flap.

## Study design and data analysis

The study will be designed as a single-arm prospective trial involving 25 eyes (of up to 25 subjects) who are presenting for LASIK retreatment. Sample size was calculated based on a nominal historical population rate of 25% ingrowth after re-lift, and an expected rate with ReSure of 5%, using an alpha of 0.05 and a power of 0.8; with these parameters a sample of 25 eyes should be sufficient to show the expected difference.

The study will involve 5 visits per eye, including a preoperative visit. Other visits will be the operative day, and 1 day, 1 week, 1 month and 3 month postoperative visits. The primary endpoint will be presence of epithelial ingrowth at 1 and 3 months after the retreatment.

NCT02952365 Document Date: September 20, 2016

Secondary endpoints will include change in refraction, best-corrected visual acuity and uncorrected visual acuity.

Inclusion criteria will be those patients who are presenting for LASIK flap re-lift and re-ablation after initial LASIK surgery. If a surgery occurs where there are intra-operative or immediate post-operative complications unrelated to the sealant the subject may be excluded from the analysis and replaced with an alternate. The data for that patient will be retained and the affected patient will be followed to monitor for adverse events, but their outcomes data would not be included in any aggregate analysis. At each visit subjects will be monitored for adverse events, whether related to the protocol regimen or not.

**Significance:** Late flap lift enhancements are associated with a higher rate of epithelial ingrowth under the flap margin. Many surgeons have stopped performing late flap lift LASIK enhancements and switched to PRK to avoid this complication. PRK over previous LASIK is associated with a prolonged visual recovery and short term ocular discomfort. If the tissue sealant is effective at preventing or lowering the rate of epithelial ingrowth under the flap, then late LASIK flap lift treatments could be offered with greater safety. This would benefit patients.

#### REFERENCES

- **1.** Mohamed TA, Hoffman RS, Fine IH, Packer M. Post-laser assisted in situ keratomileusis epithelial ingrowth and its relation to pretreatment refractive error. Cornea. 2011 May;30(5):550-2.
- 2. Levinson BA, Rapuano CJ, Cohen EJ, Hammersmith KM, Ayres BD, Laibson PR. Referrals to the Wills Eye Institute Cornea Service after laser in situ keratomileusis: reasons for patient dissatisfaction. J Cataract Refract Surg. 2008 Jan;34(1):32-9.
- 3. Caster AI, Friess DW, Schwendeman FJ. Incidence of epithelial ingrowth in primary and retreatment laser in situ keratomileusis. J Cataract Refract Surg. 2010 Jan;36(1):97-101.
- 4. Wang MY, Maloney RK. Epithelial ingrowth after laser in situ keratomileusis. Am J Ophthalmol. 2000 Jun;129(6):746-51.
- 5. Thulasi P, Kim SW, Shetty R, Randleman JB. Recalcitrant epithelial ingrowth after SMILE treated with a hydrogel ocular sealant. J Refract Surg. 2015 Dec, 31(12):847-50.
- 6. Yesillimark N, Diakonis VF, Battle JF, Yoo SH. Application of a hydrogel ocular sealant to avoid recurrence of epithelial ingrowth after LASIK enhancement. J Refract Surg. 2015 Apr:31(4):275-7.
- 7. He L. Manche EE. Fibrin glue for prevention of recurrent epithelial ingrowth under a LASIK flap with a central buttonhole defect. J Cataract Refract Surg. 2012 Oct;38(10):1857-60.
- 8. Rojas MC, Lumba JD, Manche EE. Treatment of epithelial ingrowth after laser in situ keratomileusis with mechanical debridement and flap suturing. Arch Ophthalmol. 2004 Jul;122(7):997-1001.

NCT02952365 Document Date: September 20, 2016